CLINICAL TRIAL: NCT06741501
Title: Laparoscopic Proximal Gastrectomy with "C" Single Flap Plasty Reconstruction for Upper-Third Gastric Cancer: a Randomized Clinical Trial.
Brief Title: Preliminary Efficacy Analysis of "C" Single Flap Plasty Reconstruction After Laparoscopic Proximal Gastrectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daorong Wang (Other)
Responsible Party: Sponsor-Investigator, Daorong Wang, PHD, Northern Jiangsu People's Hospital
Organization: Northern Jiangsu People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: northernjiangsu007
Record Dates: First submitted 2024-10-13; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Gastric Cancer; Reflux Esophagitis
MeSH Terms: conditions — Stomach Neoplasms; Esophagitis, Peptic

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "C" Single Flap Plasty Reconstruction (Experimental): 1. C-shaped flap creation: A 3.0 cm wide by 3.5 cm high "C"-shaped flap is marked on the anterior gastric wall, 1.5-2.5 cm distal to the stomach transection line. The flap is created by carefully separating the submucosa from the muscular propria using an electric scalpel, forming a left-opening flap. This flap will later be used to cover the anastomotic site.
  2. Esophagogastric anastomosis: The esophagus and stomach are anastomosed intracorporeally. After continuous suturing of the posterior esophageal wall to the remnant stomach, the common opening between the esophagus and the stomach is closed.
  3. Flap coverage: After anastomosis, the C-shaped flap is sutured over the anastomotic site, reinforcing it by covering both the esophageal stump and the gastric window, which helps prevent complications like leakage or reflux.
  Interventions: Procedure: "C" Single Flap Plasty Reconstruction
- Normal Reconstruction (Active Comparator): 1. Preparation of the Remnant Stomach and Esophagus: After the resection of the proximal stomach, the remaining stomach is prepared for direct anastomosis with the esophagus. The esophageal stump and gastric stump are aligned, typically without additional modifications to the gastric wall.
  2. End-to-End or End-to-Side Anastomosis: The esophagus is directly connected to the remnant stomach, either in an end-to-end or end-to-side fashion, using a stapler or manual suturing techniques.
  Interventions: Procedure: Normal Reconstruction

INTERVENTIONS:
Procedure: "C" Single Flap Plasty Reconstruction — 1. C-shaped flap creation: A 3.0 cm wide by 3.5 cm high "C"-shaped flap is marked on the anterior gastric wall, 1.5-2.5 cm distal to the stomach transection line. The flap is created by carefully separating the submucosa from the muscular propria using an electric scalpel, forming a left-opening flap. This flap will later be used to cover the anastomotic site. 2. Esophagogastric anastomosis: The esophagus and stomach are anastomosed intracorporeally. After continuous suturing of the posterior esophageal wall to the remnant stomach, the common opening between the esophagus and the stomach is closed. 3. Flap coverage: After anastomosis, the C-shaped flap is sutured over the anastomotic site, reinforcing it by covering both the esophageal stump and the gastric window, which helps prevent complications like leakage or reflux.
  Arms: "C" Single Flap Plasty Reconstruction
Procedure: Normal Reconstruction — 1. Preparation of the Remnant Stomach and Esophagus: After the resection of the proximal stomach, the remaining stomach is prepared for direct anastomosis with the esophagus. The esophageal stump and gastric stump are aligned, typically without additional modifications to the gastric wall. 2. End-to-End or End-to-Side Anastomosis: The esophagus is directly connected to the remnant stomach, either in an end-to-end or end-to-side fashion, using a stapler or manual suturing techniques.
  Arms: Normal Reconstruction

SUMMARY:
The incidence of proximal gastric cancer has increased significantly in recent years. This may be due to weight gain, alcohol consumption, gastroesophageal reflux disease (GERD), and precancerous lesions. With a deeper understanding of the pattern of lymph node metastasis and the emergence of anti-reflux procedures, proximal gastrectomy has gradually received clinical attention. For early-stage upper gastric cancer and esophagogastric combination cancer cases that are expected to have a good prognosis, the ideal surgical procedure should be to preserve the distal stomach to improve the quality of life and to choose a reasonable digestive tract reconstruction method to prevent reflux. The anti-reflux effect of various proximal gastrectomy digestive tract reconstruction methods and the advantages and disadvantages of various surgical procedures are controversial, and the recognized ideal reconstruction method has not yet been established. Therefore, we propose a reconstruction called the "C" Single Flap Plasty Reconstruction. This study aimed to investigate the efficacy and safety of proximal gastrectomy combined with "C" Single Flap Plasty Reconstruction in the treatment of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-80 years old, male or female;
2. Pathological diagnosis of preoperative endoscopic biopsy: the tumor is located in the upper 1/3 of the stomach (including the esophagogastric junction), and the clinical staging of gastric cancer： Ia and Ib (T1N0M0, T1N1M0, and T2N0M0) according to the eighth edition of the AJCC ;
3. No distant metastasis was observed on preoperative chest radiograph, abdominal ultrasound, or upper abdominal CT;
4. ASA grade 1-3;
5. Patients without contraindications to surgery;
6. Patients and their families voluntarily signed the informed consent form and participated in the study;

Exclusion Criteria:

1. Patients diagnosed with primary tumors or distant metastasis;
2. Patients whose tumor is located in the greater curvature side of the stomach;
3. Patients with coagulation dysfunction that could not be corrected;
4. Patients who were diagnosed with viral hepatitis and cirrhosis;
5. Patients who were diagnosed with diabetes mellitus, uncontrolled or controlled with insulin;
6. Patients with organ failure such as heart, lung, liver, brain, and kidney failure;
7. Patients with ascites or cachexia preoperatively in poor general conditions;
8. Patients diagnosed with immunodeficiency, immunosuppression, or autoimmune diseases (such as allogeneic bone marrow transplant, immunosuppressive drugs, SLE, etc.).
9. Patients refusing to sign the informed consent of the study;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
incidence of reflux esophagitis | 6 months after surgery
  The percentage (%) of patients developing postoperative reflux esophagitis after surgery in each group.

SECONDARY OUTCOMES:
incidence of anastomotic leakage | 30 days after surgery
  The percentage (%) of patients developing postoperative anastomotic leakage after surgery in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No